CLINICAL TRIAL: NCT03401099
Title: Cryoballoon Pulmonary Vein Isolation as First Line Treatment for Typical Atrial Flutter
Brief Title: Cryoballoon Ablation as First Line Treatment of Atrial Flutter
Acronym: CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Medtronic International Trading Sarl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1153
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Atrial Flutter Typical
Keywords: Radiofrequency ablation; Cavo-tricuspid isthmus; Pulmonary Vein Isolation; Cryoballoon ablation

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 into two groups to receive either of the two treatments.
Who Masked: Outcomes Assessor
Masking Description: Blinded outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation of CTI (Active Comparator): Radiofrequency ablation of CTI (cavo-tricuspid isthmus), which is the 'conventional' treatment of atrial flutter
  Interventions: Procedure: Radiofrequency ablation of CTI
- Cryoballoon PVI (Active Comparator): Cryoballoon PVI (Pulmonary Vein Isolation), which is the 'novel treatment'
  Interventions: Procedure: Cryoballoon PVI

INTERVENTIONS:
Procedure: Radiofrequency ablation of CTI — Delivery of radiofrequency energy to the cavotricuspid isthmus (region of right atrial tissue between the tricuspid annulus and the inferior vena cava) until bidirectional block is achieved
  Other Names: CTI ablation
  Arms: Radiofrequency ablation of CTI
Procedure: Cryoballoon PVI — Cryoballoon application to the pulmonary veins aiming for Pulmonary Vein Isolation
  Other Names: Cryoablation Pulmonary Vein Isolation
  Arms: Cryoballoon PVI

SUMMARY:
Current guidelines recommend radiofrequency catheter ablation of the cavotricuspid isthmus as treatment for symptomatic/drug-refractory atrial flutter, in spite of the fact that recurrences of flutter and incidence of post-ablation atrial fibrillation are common.

In this study, the investigators assess the hypothesis that the use of cryoballoon Pulmonary Vein Isolation ('novel' treatment) to achieve the electrical disconnection between the pulmonary veins and the heart will lead to higher rates of freedom from abnormal heart rhythms (atrial flutter, atrial fibrillation, or atrial tachycardia) and more improved quality of life than treatment using heat energy (radiofrequency ablation) directed at the cavotricuspid isthmus ('conventional treatment').

DETAILED DESCRIPTION:
Atrial flutter and atrial fibrillation are believed to share the same initiating triggers in the form of pulmonary vein ectopy. Cavo-tricuspid isthmus-dependent atrial flutter almost always results from short bursts of antecedent atrial fibrillation. Radiofrequency (RF) ablation of the cavo-tricuspid isthmus (CTI) is the current accepted first-line treatment for atrial flutter, although post-ablation atrial fibrillation commonly occurs, even in the absence of pre-existing atrial fibrillation.

Cryoballoon Pulmonary Vein Isolation (PVI) has become an established treatment for atrial fibrillation. In patients with both atrial flutter and fibrillation, PVI alone has been shown to control both types of atrial arrhythmia, with no benefit derived from supplemental RF CTI ablation.

This study aims to demonstrate that standalone cryoballoon PVI for typical atrial flutter without RF CTI ablation will lead to a significant difference in preventing recurrence of atrial arrhythmia compared to radiofrequency ablation of the CTI, and should be offered as first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years
* 2. Patients referred for catheter ablation for typical atrial flutter. The atrial flutter may be either persistent or paroxysmal, with at least one episode having been documented on 12-lead ECG. In the view of the treating physician, the ECG morphology should be compatible with a CTI-dependent circuit, either counterclockwise or clockwise.

Exclusion Criteria:

* 1. Any evidence of previously documented atrial fibrillation
* 2. Previous cavo-tricuspid isthmus ablation or atrial fibrillation ablation
* 3. Atrial flutter documented solely on Ambulatory monitoring
* 4. Atrial flutter morphology on ECG suggestive of a left atrial flutter
* 5. History of atrial flutter with 1:1 atrioventricular conduction and haemodynamic compromise
* 6. Indwelling atrial-septal defect occluder device, or any anatomical reason that precludes left atrial access
* 7. Left atrial diameter (PLAX M-mode) >5.5 cm
* 8. Severe left ventricular dysfunction (LV ejection fraction < 30% on Echocardiography)
* 9. Recent stroke/transient ischaemic attack within 3 months
* 10. Inability or unwillingness to take oral anticoagulant treatment
* 11. Morbid obesity (Body Mass Index ≥40)
* 12. Extreme frailty (A score of 7,8 or worse on the Clinical Frailty Scale)
* 13. Implanted metal prosthetic valve(s) in mitral position
* 14. Indwelling cardiac resynchronisation therapy device, pacemaker or implantable cardioverter defibrillator
* 15. Advanced Renal dysfunction (eGFR<30 ml/min)
* 16. Pregnancy
* 17. Severe valvular heart disease of any kind as assessed by the investigator
* 18. Previous valve replacement surgery or other prosthetic heart valve

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence of sustained, symptomatic supraventricular arrhythmia (Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia) following a blanking period of 4 weeks after a single ablation procedure | After 4 weeks of ablation treatment (blanking period) up to 12 months of follow up
  'Sustained' is defined as lasting >30 seconds. 'Symptomatic' is defined as acute onset awareness of palpitations, breathlessness, dizziness, fatigue or chest pain associated with patient activation of the loop recorder.

SECONDARY OUTCOMES:
Time to first symptomatic or asymptomatic Atrial Fibrillation lasting ≥2 min | After 4 weeks of ablation treatment (blanking period) up to 12 months of follow up
  How long it takes until first occurrence of atrial fibrillation (associated with symptoms or no symptoms) lasting 2 or more minutes after blanking period. Two minutes is the minimum duration detectable by the loop recorder
Total Burden of Atrial fibrillation over 12 months | After 4 weeks of ablation treatment (blanking period) up to 12 months of follow up
  The total occurrence of atrial fibrillation recorded by the loop recorder (symptomatic or asymptomatic) during the follow-up period
Time to first symptomatic or asymptomatic atrial flutter/atrial tachycardia | After 4 weeks of ablation treatment (blanking period) up to 12 months of follow up
  Occurrence of atrial flutter/atrial tachycardia with/without symptoms following the blanking period
Incidence of any significant arrhythmia | After first ablation procedure, through study completion, an average of 12 months
  Incidence of any arrhythmia requiring medical visit to primary or secondary care, or hospitalisation, or leading to death
Total burden of abnormal heart rhythm measured by the implantable loop recorder | After first ablation procedure through study completion or time of intervention, whichever comes first, assessed up to 12 months
  Total arrhythmic burden up to end of follow up or up to time of intervention (either cardioversion or ablation), whichever comes first.
Incidence of repeat electrophysiological interventional procedure (repeat catheter ablation, or DCCV) over the follow-up period. | After 4 weeks of ablation treatment (blanking period) up to 12 months of follow up
  Occurrence of repeat ablations/cardioversion
Incidence of procedural complications | During and after ablation procedure, through study completion, an average of 12 months
  Composite of cardiac tamponade requiring drainage, persistent phrenic nerve palsy lasting >24 hours, serious vascular complications requiring intervention or delaying discharge, stroke/transient ischaemic attack, requirement for a permanent pacemaker, atrio-esophageal fistula, or death
Incidence of all-cause hospitalisations | After first ablation procedure, through study completion, an average of 12 months
  Any hospital admission post-ablation
Quality of Life questionnaire | At baseline and at 12 months
  Quality of life as assessed by the standard EuroQol Group's 5-dimensional questionnaire. This comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the visual analogue scale. The single digits for the five dimensions will be combined into a 5-digit number that describes the patient's health state.
Procedural duration | Only during the first ablation procedure
  Duration of ablation measured in minutes for either treatment
Total Fluoroscopy times | Only during the first ablation procedure
  The total time in minutes during which patient will be exposed to radiation under each of the two treatment techniques

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MBBS MD FRCP, Study Chair — Liverpool Heart and Chest Hospital
Locations (10):
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Inselspital Bern, Bern
- United Kingdom (8):
  - Royal Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Manchester University NHS Foundation Trust, Wythenshawe Hospital, Manchester
  - South Tees Hospitals NHS Foundation Trust, James Cook University Hospital, Middlesbrough
  - The Newcastle Upon Tyne Hospital NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, John Radcliffe Hospital, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant Data with other researchers.
  Supporting information that will be shared are only:
  Study Protocol, Statistical Analysis Plan (SAP), and Clinical Study Report (CSR)
  Data will be available after about 6 months for about 5 years.
  Criteria for which Individual Participant Data and any additional supporting information will be shared, including with whom, for what types of analyses, and by what mechanism:
  These will be shared with research co-workers, for results, statistical analysis and conclusions. Communication of anonymized data will be done via secure mails and emails.

REFERENCES:
- [Background] Wazni O, Marrouche NF, Martin DO, Gillinov AM, Saliba W, Saad E, Klein A, Bhargava M, Bash D, Schweikert R, Erciyes D, Abdul-Karim A, Brachman J, Gunther J, Pisano E, Potenza D, Fanelli R, Natale A. Randomized study comparing combined pulmonary vein-left atrial junction disconnection and cavotricuspid isthmus ablation versus pulmonary vein-left atrial junction disconnection alone in patients presenting with typical atrial flutter and atrial fibrillation. Circulation. 2003 Nov 18;108(20):2479-83. doi: 10.1161/01.CIR.0000101684.88679.AB. Epub 2003 Nov 10. PMID 14610012
- [Background] Schneider R, Lauschke J, Tischer T, Schneider C, Voss W, Moehlenkamp F, Glass A, Diedrich D, Bansch D. Pulmonary vein triggers play an important role in the initiation of atrial flutter: Initial results from the prospective randomized Atrial Fibrillation Ablation in Atrial Flutter (Triple A) trial. Heart Rhythm. 2015 May;12(5):865-71. doi: 10.1016/j.hrthm.2015.01.040. Epub 2015 Jan 28. PMID 25638698
- [Background] De Bortoli A, Shi LB, Ohm OJ, Hoff PI, Schuster P, Solheim E, Chen J. Incidence and clinical predictors of subsequent atrial fibrillation requiring additional ablation after cavotricuspid isthmus ablation for typical atrial flutter. Scand Cardiovasc J. 2017 Jun;51(3):123-128. doi: 10.1080/14017431.2017.1304570. Epub 2017 Mar 23. PMID 28335638
- [Derived] Gupta D, Ding WY, Calvert P, Williams E, Das M, Tovmassian L, Tayebjee MH, Haywood G, Martin CA, Rajappan K, Bates MGD, Temple IP, Reichlin T, Chen Z, Balasubramaniam RN, Ronayne C, Clarkson N, Morgan M, Barton J, Kemp I, Mahida S, Sticherling C. Cryoballoon Pulmonary Vein Isolation as First-Line Treatment for Typical Atrial Flutter. Heart. 2023 Feb 14;109(5):364-371. doi: 10.1136/heartjnl-2022-321729. PMID 36396438
- [Derived] Ding WY, Williams E, Das M, Tovmassian L, Tayebjee M, Haywood G, Martin C, Rajappan K, Bates M, Temple IP, Reichlin T, Chen Z, Balasubramaniam R, Ronayne C, Clarkson N, Mahida S, Sticherling C, Gupta D. Cryoballoon pulmonary vein isolation as first line treatment for typical atrial flutter (CRAFT): study protocol for a randomised controlled trial. J Interv Card Electrophysiol. 2021 Apr;60(3):427-432. doi: 10.1007/s10840-020-00746-6. Epub 2020 May 8. PMID 32385774